CLINICAL TRIAL: NCT01254253
Title: Multimodality Imaging Evaluation of Functional and Clinical Benefits of Percutaneous Coronary Intervention in Patients With Chronic Total Occlusion Lesion
Brief Title: Functional and Clinical Benefits of PCI in Patients With CTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFFECT
Record Dates: First submitted 2010-12-01; First posted 2010-12-06 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Heart Function; Quality of Life
Keywords: percutaneous coronary intervention; chronic total occlusion; coronary angiography; single photon emission CT; Multislice coronary CT angiography
MeSH Terms: interventions — Percutaneous Coronary Intervention; Treatment Outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group a (Experimental): no severe cardiac perfusion defects
  Interventions: Device: Percutaneous coronary intervention, PCI
- Gooup b (Experimental): reversible cardiac perfusion defects
  Interventions: Device: Percutaneous coronary intervention, PCI
- Group c (Experimental): irreversible cardiac perfusion defects
  Interventions: Device: Percutaneous coronary intervention, PCI

INTERVENTIONS:
Device: Percutaneous coronary intervention, PCI — PCI was performed using standard techniques for CTO.
  Other Names: Effect; Xijing Hospital, Fourth Military Medical University

SUMMARY:
The purpose of this study is to compare the diagnostic accuracy of hybrid imaging combining CTCA with low-dose stress-only SPECT vs. coronary angiography for detecting haemodynamic relevant coronary lesions; and second to determine the effects of PCI on cardiac perfusion, cardiac function and quality of life in patients with CTO lesion in left anterior descending (LAD) coronary artery.

DETAILED DESCRIPTION:
Noninvasive imaging modalities have shown high diagnostic accuracy in the detection of coronary artery lesions, and for the estimation of their hemodynamic relevance.Thus, noninvasive assessment of myocardial perfusion defects may be preferred for patients with chronic total occlusion (CTO).

In particular, myocardial perfusion is measured with single photon emission CT (SPECT).Multislice coronary CT angiography (CCTA) with dual-source scanners reveals the anatomic location of coronary artery disease (CAD). These two techniques assess distinct aspects of heart morphology and function parameters of the heart, and should therefore be regarded as complementary rather than competing methods.Taking this into consideration, decisions regarding whether invasive revascularization therapy is adequate or not and which strategy is the best for long-term survival cannot be supported by anatomic information alone. Therefore, noninvasive complementary imaging of structure and perfusion, in conjunction with three-dimensional (3D) image fusion, has emerged as a technique for reliable allocation of perfusion defects to their supplying coronary artery.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for enrolment in this study if coronary angiography showed a CTO (at least for 3 months and confirmed by angiography and/or history of earlier MI).

Exclusion Criteria:

* Hypersensitivity to iodinated contrast agent, cardiomyopathy, non-sinus rhythm, severe valvular heart disease, NYHA functional class IV heart failure at baseline, previous coronary bypass surgery, renal insufficiency, severe lung and liver disease or cancer.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 2year

SECONDARY OUTCOMES:
cardiac death | 2year
Non-fatal myocardial infarction | 2 year
Target lesion revascularization | 2 year
Angina pectoris score index | 2 year
Six-minute walk distance | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Feng Cao, MD, PhD, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Fourth Military Medical University, Xi'an, Shaanxi, China